CLINICAL TRIAL: NCT00396630
Title: A Phase IIIb, Randomized, Double-Blind, Placebo-Controlled Study to Explore the Existence of Horizontal Transmission of the RIX4414 Vaccine Strain Between Twins Within a Family.
Brief Title: A Study to Explore the Existence of Horizontal Transmission of the RIX4414 Vaccine Strain Between Twins Within a Family.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 106260
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Results first posted 2009-03-13 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2017-11

CONDITIONS: Infections, Rotavirus
Keywords: Transmission; Gastroenteritis; Shedding; rotavirus; HRV vaccine
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rotarix Group (Experimental): All subjects received 2 oral doses of Rotarix vaccine at Day 0 (Visit 1) and Week 7 (Visit 2).
  Subjects aged less than 6 months at Visit 3 received one complimentary Rotarix vaccine dose at Week 13 (Visit 3).
  Interventions: Biological: Rotarix
- Placebo Group (Placebo Comparator): All subjects received 2 oral doses of placebo at Day 0 (Visit 1) and Week 7 (Visit 2).
  Subjects aged less than 6 months at Visit 3 received one complimentary Rotarix vaccine dose at Week 13 (Visit 3).
  Interventions: Biological: Rotarix; Biological: Placebo

INTERVENTIONS:
Biological: Rotarix — Two-dose oral vaccination.
Biological: Placebo — Two-dose oral administration.
  Arms: Placebo Group

SUMMARY:
The aim of this study is to explore horizontal transmission of the HRV (Human Rotavirus) vaccine strain within a family from the twin vaccinated with Rotarix to the twin receiving placebo. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This is a Phase 3b study. Three doses of Infanrix® hexa will be administered to all subjects at the discretion of the investigator.

One complimentary dose of Rotarix will be administered to all infants enrolled in this study (both study groups) who are aged less than 6 months at Visit 3 (Week 13) as a benefit to the placebo group for participation in the study.

The study will be conducted in a double-blind manner with respect to Rotarix and placebo administered at Visit 1 and Visit 2. The parents/guardians of the subjects will know that within each pair of twins, one subject will receive the Rotarix vaccine and one subject will receive the placebo.

The study will be open label with respect to administration of the Rotarix vaccine dose given at Visit 3 to all subjects in each group who are aged less than 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a live twin living in the same household who is also enrolled in this study.
* Born after a gestation period of ≥32 weeks,
* Discharged from hospital neonatal care stay,
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 14 weeks of age at the time of the first study vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parent or guardian of the subjects.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Any clinically significant history of chronic gastrointestinal disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Contact with an immunosuppressed individual.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants since birth.
* Gastroenteritis within 7 days preceding the first study vaccine administration.
* Documented HIV-positive subject.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2007-01-23 (Actual); Primary Completion 2008-01-23 (Actual); Study Completion 2008-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Rivera L, Pena LM, Stainier I, Gillard P, Cheuvart B, Smolenov I, Ortega-Barria E, Han HH. Horizontal transmission of a human rotavirus vaccine strain--a randomized, placebo-controlled study in twins. Vaccine. 2011 Nov 28;29(51):9508-13. doi: 10.1016/j.vaccine.2011.10.015. Epub 2011 Oct 18. PMID 22008819
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Within each pair of twins enrolled in the study, one subject was assigned to the Rotarix Group and one to the Placebo Group.
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 100 | 100
Completed | 95 (Completed Visit 4 (Week 17).) | 95 (Completed Visit 4 (Week 17).)
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not vaccinated at Visit 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.2 (1.80) | 8.2 (1.80) | 8.2 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 49 | 105
  Male | 44 | 51 | 95

OUTCOME MEASURES:

1. Primary Outcome: Presence of Rotavirus Vaccine Strain in Any Stool Sample From Twin Receiving Placebo.
Description: Number of subjects in the Placebo Group with rotavirus vaccine strain in at least one stool sample.
Time Frame: On the day of each vaccine/placebo dose, then three times weekly for 6 consecutive weeks starting after each vaccine/placebo dose and on the day of Visit 3.
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Placebo Group
Number analyzed (Participants) | 80
subjects | 15

2. Secondary Outcome: Duration of Human Rotavirus (HRV) Shedding Per Study Group.
Description: Duration of shedding in the Placebo Group= number of days between first and last stool sample positive (+) for rotavirus (RV) antigen and in the Rotarix Group= number of days between the day of vaccination and the date of last stool sample + for RV antigen.
Time Frame: From Day 0 up to Week 13.
Population: The analysis was performed on the According To Protocol analysis for immunogenicity, on the twins whose placebo recipient had at least one stool sample positive for the rotavirus strain.
Measure: Median (Inter-Quartile Range); unit: Number of days
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 15 | 15
Number of days
  After Dose 1 (n=11, 9) | 17 [11 to 19] | 7 [3 to 13]
  After Dose 2 (n=9, 7) | 13 [5 to 17] | 1 [1 to 1]

3. Secondary Outcome: Number of Genetic Variation Differences Detected by Sequencing of Genomic Mutations in the HRV Vaccine Strain After Transmission.
Description: Dissimilar amino acid substitutions in the HRV vaccine strain isolated from the twin receiving placebo, when compared to the genetic variation of HRV vaccine strain isolated from the Rotarix vaccine recipients, were counted as genetic variation differences.
Time Frame: During the entire study period (up to Visit 4, Week 17).
Population: The analysis was performed on the According To Protocol analysis for immunogenicity, on the twins who received placebo and those who received Rotarix vaccine, in case of transmission.
Measure: Number; unit: Genetic variation difference
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 15 | 15
Genetic variation difference | 0 | 0

4. Secondary Outcome: Live Viral Vaccine Load in the Stool of the Twin Receiving Placebo in Case of Transmission.
Description: Number of subjects in the Placebo Group with live virus identified in at least one stool sample in case of transmission.
Time Frame: During the entire study period (up to Visit 4, Week 17).
Population: The analysis was performed on the According To Protocol analysis for immunogenicity, on the twins who received placebo in case of transmission.
Measure: Number; unit: Subjects
Arm/Group | Placebo Group
Number analyzed (Participants) | 15
Subjects | 3

5. Secondary Outcome: Anti-rotavirus Immunoglobulin A (IgA) Antibody Seroconversion.
Description: Number of initially seronegative subjects with anti-rotavirus IgA antibody concentration ≥ 20 Units/milliliter (U/mL), 1 month after the second dose.
Time Frame: At Visit 3 (Week 13).
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 80 | 80
subjects | 50 | 17

6. Secondary Outcome: Anti-rotavirus IgA Antibody Concentration.
Description: Anti-rotavirus IgA antibody concentrations are given as geometric mean concentrations (GMC) with 95% Confidence Intervals.
Time Frame: At Visit 3 (Week 13).
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 80 | 80
U/mL | 78.6 [50.6 to 122.2] | 20.5 [14.5 to 28.9]

7. Secondary Outcome: Number of Subjects With Gastroenteritis (GE) and Rotavirus Gastroenteritis (RV GE) Episodes.
Description: GE episodes were defined as diarrhea (passage of three or more looser than normal stools within a day) with or without vomiting.
  RV GE episodes were defined as GE episodes for which the stool sample temporally closest to the onset day of the GE episode was positive for rotavirus by Enzyme Linked Immunosorbent Assay (ELISA).
Time Frame: Until Visit 4 (Week 17) for GE and until Visit 3 (Week 13) for RV GE.
Population: The analyses were performed on the Total Vaccinated Cohort
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 100 | 100
subjects
  GE episodes | 32 | 31
  RV GE episodes | 10 | 6

8. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 31 days after any doses.
Population: The analyses were performed on the Total Vaccinated Cohort
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 100 | 100
subjects | 69 | 71

9. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: A serious adverse event (SAE) is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Up to Visit 4.
Population: The analyses were performed on the Total Vaccinated Cohort
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 100 | 100
subjects | 5 | 6

ADVERSE EVENTS:
Arm/Group | Rotarix Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 5/100 | 6/100
Other Adverse Events (participants affected / at risk) | 69/100 | 71/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=100) | Placebo Group (N=100)
Bronchiolitis (Infections and infestations) | 3 | 3
Gastroenteritis (Infections and infestations) | 2 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=100) | Placebo Group (N=100)
Nasopharyngitis (Infections and infestations) | 49 | 49
Pyrexia (General disorders) | 32 | 32
Irritability (General disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.